CLINICAL TRIAL: NCT02736318
Title: Treatment of Osteochondral Lesion of Talus With Processed Osteochondral Allograft
Brief Title: OD-PHOENIX in Talus Osteochondral Lesion
Acronym: TBF3
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBFLab
Record Dates: First submitted 2016-04-01; First posted 2016-04-13 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Talus Osteochondral Defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- processed osteochondral allograft (Experimental): Implantation of 1 to 3 osteochondral products in osteochondral lesion of talus.
  Interventions: Biological: OD-PHOENIX

INTERVENTIONS:
Biological: OD-PHOENIX — Decellularized, freeze-dried, irradiated osteochondral allograft
  Other Names: Osteochondral allograft

SUMMARY:
Treatment of osteochondral lesion of Talus with a devitalized viro-inativated sterile osteochondral graft. To avoid having to harvest autograft material from the knee, a processed allogeneic osteochondral can be used instead autograft. The surgical technique is to implant in the osteochondral defect one to three products in the defect.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18 and 50
* Isolated osteochondral lesion of the talus due to trauma (fracture) or osteochondritis dissecans
* Osteochondral lesion > Anderson Grade I (MRI)
* 1 to 3 cm2 lesion
* Presence of disabling and clinically meaningful symptoms (subjective OMAS < 50)
* Patient who has been treated previously for this lesion, except if this treatment consisted of autologous osteochondral grafting
* No significant obesity (BMI < 30)
* Patient able to understand, sign and date the informed consent form
* Patient affiliated with a national health insurance system or who is the beneficiary of such as system
* Women of childbearing age may not be included in the clinical trial unless their pregnancy test is negative. If this test is negative, they will be asked to use an effective birth control method during the entire the study.

Exclusion Criteria:

* Pregnant or breast feeding women: Women of childbearing age will be asked to undergo a pregnancy test before being enrolled into the study and to use an effective birth control method.
* Previous mosaicplasty treatment of this lesion
* Fracture or bone defect or subchondral lesion without cartilage involvement, untreated osteonecrosis, collapse of talar dome
* Presence of osteoarthritis, rheumatoid arthritis, excessive hindfoot deformity or any other condition of the talocural joint that, in the surgeon's opinion, is likely to compromise the allograft's outcome
* Excessive laxity or recurrent instability that could affect the score evaluation
* Presence of an ulcerative disease, heavy smoking, tuberculosis, chronic psychiatric disorder or disease requiring long-term treatment with a medication that would affect bone or joint metabolism
* Persons with cancer or a history of cancer
* Persons deprived of their freedom by a judicial or administrative decision
* Adults subject to legal protection measures or who are unable to provide their consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Determine the improvement in ankle function based on the OMAS at 24 months | 3 months, 6 months, 12 months, 18 months, 24 months
  questionnaire

SECONDARY OUTCOMES:
Clinical and functional improvement of the ankle by AOFAS score | 3 months, 6 months, 12 months, 18 months,24 months
  questionnaire and clinical evaluation
Impairment improvement by FASS ( foot and ankle severity score) | 3 months, 6 months, 12 months, 18 months,24 months
  questionnaire
Evaluate osteochondral graft integration with imaging | 12 months, 18 months, 24 monts
  - CT-scan at 12 months, MRI 18- 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- AZ Monica, Antwerp, Belgium
- Poriya Medical Center, Tiberias, Israel

IPD SHARING:
Plan to Share IPD: Undecided